CLINICAL TRIAL: NCT02139878
Title: Short-term Health Effects of Wild Blueberry Juice Consumption
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Prince Edward Island (Other)
Responsible Party: Principal Investigator, Kim Stote, Research Chair of Nutrisciences and Health, University of Prince Edward Island
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Other
Other Study IDs: UPEI HS 01
Record Dates: First submitted 2014-05-04; First posted 2014-05-15 (Estimated); Results first posted 2017-02-17 (Actual); Last update posted 2017-03-28 (Actual); Status verified 2016-12

CONDITIONS: Pre-diabetes
MeSH Terms: conditions — Glucose Intolerance

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Wild blueberry juice (Experimental): 240 ml wild blueberry juice
  Interventions: Other: Wild blueberry juice
- Placebo wild blueberry juice (Placebo Comparator): 240 ml placebo wild blueberry juice
  Interventions: Other: Placebo wild blueberry juice

INTERVENTIONS:
Other: Wild blueberry juice
  Arms: Wild blueberry juice
Other: Placebo wild blueberry juice
  Arms: Placebo wild blueberry juice

SUMMARY:
Researchers at the University of Prince Edward Island want to learn about the health effects of wild blueberry juice.

ELIGIBILITY:
Inclusion Criteria:

* Healthy individuals at risk for type 2 diabetes

Exclusion Criteria:

* have a body mass index of less than 20 and greater than 45 kg/m2.
* are less than 21 and greater than 65 years old at beginning of study
* have smoked or used tobacco within 6 months prior to the start of the study
* are pregnant, plan to become pregnant or become pregnant during the study
* have a history or presence of kidney disease, liver disease, certain cancers, gastrointestinal, other metabolic diseases, or malabsorption syndromes
* have type 2 diabetes and need to use oral diabetic drugs or insulin
* have an allergy or adverse reaction to blueberries

Ages: 25 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2014-05; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Katherine Gottschall-Pass, PhD, RD, Principal Investigator — University of Prince Edward Island
Locations (1):
- University of Prince Edward Island, Health Sciences, Charlottetown, Prince Edward Island, Canada

REFERENCES:
- [Derived] Stote KS, Sweeney MI, Kean T, Baer DJ, Novotny JA, Shakerley NL, Chandrasekaran A, Carrico PM, Melendez JA, Gottschall-Pass KT. The effects of 100% wild blueberry (Vaccinium angustifolium) juice consumption on cardiometablic biomarkers: a randomized, placebo-controlled, crossover trial in adults with increased risk for type 2 diabetes. BMC Nutr. 2017 May 25;3:45. doi: 10.1186/s40795-017-0164-0. eCollection 2017. PMID 32153825

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 74 individuals were screened for eligibility from the greater Charlottetown, Prince Edward Island, Canada area from March 2014 to May 2014.
Pre-assignment Details: 20 of the 74 participants were randomized. Of those not randomized, 49 did not meet the inclusion criteria and 5 declined to participate.
Groups:
- Wild Blueberry Juice First, Then Placebo: 240 ml Wild Blueberry Juice daily first in intervention period and 240 ml Placebo beverage daily in second intervention period (after washout period)
- Placebo First, Then Wild Blueberry Juice: 240 ml Placebo beverage daily in first intervention period and 240 ml Wild Blueberry Juice daily in second intervention period (after washout period).
Period: First Intervention (7 Days)
Arm/Group | Wild Blueberry Juice First, Then Placebo | Placebo First, Then Wild Blueberry Juice
Started | 10 | 10
Completed | 9 | 10
Not Completed | 1 | 0
Period: Washout Period (8 Days)
Arm/Group | Wild Blueberry Juice First, Then Placebo | Placebo First, Then Wild Blueberry Juice
Started | 9 | 10
Completed | 9 | 10
Not Completed | 0 | 0
Period: Second Intervention (7 Days)
Arm/Group | Wild Blueberry Juice First, Then Placebo | Placebo First, Then Wild Blueberry Juice
Started | 9 | 10
Completed | 9 | 10
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Entire Study Population: Includes groups randomized to receive Wild Blueberry Juice first and Placebo first
Arm/Group | Entire Study Population
Number analyzed (Participants) | 19
Age, Continuous [Mean (Standard Deviation); unit: years] | 53 (6.3)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: 1 participant was randomized but did not start the study
  Participants
    Female | 19
    Male | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 19
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  Canada | 19

OUTCOME MEASURES:

1. Primary Outcome: Blood Pressure
Description: Systolic blood pressure
Time Frame: Up to 4 weeks
Measure: Mean (Standard Error); unit: mm Hg
Groups:
- Placebo: 240 ml placebo beverage
Arm/Group | Wild Blueberry Juice | Placebo
Number analyzed (Participants) | 19 | 19
mm Hg | 116.0 (2.2) | 120.8 (2.2)
Statistical Analysis 1: Comparison: Wild Blueberry Juice vs Placebo; Test type: Superiority or Other; p = 0.088, ANCOVA

2. Secondary Outcome: Glucose
Description: Plasma blood glucose concentrations
Time Frame: Up to 4 weeks
Measure: Mean (Standard Error); unit: mmol/L
Arm/Group | Wild Blueberry Juice | Placebo
Number analyzed (Participants) | 19 | 19
mmol/L | 5.3 (0.1) | 5.4 (0.1)
Statistical Analysis 1: Comparison: Wild Blueberry Juice vs Placebo; Test type: Superiority or Other; p = 0.980, ANCOVA

ADVERSE EVENTS:
Groups:
- Wild Blueberry Juice: 240 ml Wild Blueberry Juice daily in either first intervention period or second intervention period
- Placebo: 240 ml Placebo beverage daily in either the first intervention period or second intervention period
Arm/Group | Wild Blueberry Juice | Placebo
Serious Adverse Events (participants affected / at risk) | 0/19 | 0/19
Other Adverse Events (participants affected / at risk) | 0/19 | 0/19

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No